CLINICAL TRIAL: NCT02253394
Title: The Combination Ambrisentan Plus Spironolactone in Pulmonary Arterial Hypertension Study (The CAPS-PAH Study)
Brief Title: The Combination Ambrisentan Plus Spironolactone in Pulmonary Arterial Hypertension Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Bradley Maron, MD, Instructor in Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CAPS_PAH
Record Dates: First submitted 2014-09-17; First posted 2014-10-01 (Estimated); Results first posted 2019-11-15 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial Hypertension (PAH); Ambrisentan; Spironolactone; Selective Endothelin A (ETA) inhibition; Aldosterone antagonism; Cardiac output (CO); Right ventricular (RV) function; Heart failure; Quality of life; Pro-inflammatory cytokine; Interleukin-6 (IL-6); Troponin-I; N-terminal pro-brain natriuretic peptide (NT-BNP); Collagen metabolism; N-terminal procollagen type I; Collagen III; Echocardiography; WHO Functional Class; Cardiopulmonary Exercise Test with Innocor; Peak oxygen consumption (pVO2); Liver function markers (AST/ALT); Renal function markers (creatinine and potassium)
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Inhibition, Psychological; Heart Failure | interventions — ambrisentan; Spironolactone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- AMB + Spiro, Cardiopulmonary fitness (Active Comparator): Ambrisentan 5 or 10 mg every day (QD) Spironolactone 50 mg QD
  Interventions: Drug: Ambrisentan plus Spironolactone
- Placebo Cardiopulmonary fitness (Placebo Comparator): Placebo mimics spironolactone 50 mg and will be taken QD
  Interventions: Drug: Ambrisentan plus Placebo

INTERVENTIONS:
Drug: Ambrisentan plus Spironolactone — Cardiopulmonary fitness
  Other Names: Letairis plus Aldactone
  Arms: AMB + Spiro, Cardiopulmonary fitness
Drug: Ambrisentan plus Placebo — Placebo is a sugar pill manufactured to resemble spironolactone 50 mg Cardiopulmonary fitness
  Other Names: Letairis
  Arms: Placebo Cardiopulmonary fitness

SUMMARY:
The purpose of this study is to find out if spironolactone added to ambrisentan for Pulmonary Arterial Hypertension (PAH) will increase exercise capacity. We also want to find out if spironolactone and ambrisentan effect the cardiac output (amount of blood the heart pumps every minute), right ventricle function and quality of life.

DETAILED DESCRIPTION:
A prospective, double blind, placebo-controlled clinical study involving 30 patients with World Health Organization (WHO) Group 1 pulmonary arterial hypertension being treated with ambrisentan randomized to receive placebo or spironolactone (50 mg/d) for 90 days using a cross-over trial design.

Eligible participants will be randomized to receive placebo or spironolactone (50 mg/d) for 90 days (Phase I). At the completion of Phase I, participants will undergo repeat end-point assessment followed by a 21-day drug washout period. Then, the 90 day crossover phase of the trial will occur (Phase II), in which participants randomized to placebo in Phase I will be treated with spironolactone (50 mg/d) in Phase II and vice versa. At the conclusion of Phase II, end-point measures are reassessed.

Spironolactone is a diuretic used in treatment of PAH patients. Spironolactone is usually added to medical treatment when doses of Lasix/Torsemide are increased and patients are at risk for hypokalemia.

Study procedures being done for this research study are the standard procedures performed on all PAH patients when they are in clinic for follow-up except for the Cardiopulmonary Exercise Test (CPET) with Innocor.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily gives informed consent to participate in the study.
2. Right heart catheterization demonstrating conventional mean pulmonary artery pressure (mPAP) >25, pulmonary vascular resistance (PVR) >3.0 Wood Units, pulmonary capillary wedge pressure (PCWP) <16 mmHg within two years of enrollment
3. Subject is 18 years of age or older at Screening.
4. Diagnosis of symptomatic idiopathic or heritable PAH, PAH associated with Connective Tissue Disease (CTD), PAH associated with repaired/unrepaired congenital systemic-to-pulmonary shunt, Portopulmonary hypertension or PAH associated with HIV infection.
5. New York Heart Association Functional Class II or III
6. Stable therapy with ambrisentan 5 or 10 mg every day for > 90 days.
7. Baseline 6-Minute Walk Distance 50-450m

Exclusion Criteria:

1. Substantial Primary Lung disease

   * forced expiratory volume at one second (FEV-1)/forced vital capacity (FVC) <0.6 and FEV-1 <70% predicted
   * diffusing capacity of lung for carbon monoxide (DLCO) <30% predicted
   * Pulmonary fibrosis
2. Left ventricular ejection fraction < 50%
3. Pulmonary capillary wedge pressure > 16 mm Hg
4. Aortic valve disease
5. Ischemic heart disease
6. Systemic hypotension (SBP <90 mm Hg)
7. Co-existing treatment with other endothelin receptor antagonists or prostacyclin analogues
8. New York Heart Association Functional Class IV
9. Chronic thromboembolic pulmonary hypertension
10. Known or suspected pulmonary veno-occlusive disease
11. Serum creatinine >2.0 mg/dL in women, Serum creatinine >2.5 mg/dL in men
12. Baseline serum potassium >5.0 milliequivalent (mEq)/L
13. Participation in ongoing drug/intervention-based clinical trial
14. Pregnancy
15. Unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Maron, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- AMB + Spiro First, Then Placebo, Cardiopulmonary Fitness: Ambrisentan 5 or 10 mg every day (QD) plus Spironolactone 50 mg QD FIRST, then placebo
- AMB + Placebo First, Then Spironolactone: Ambrisentan 5 or 10 mg every day (QD) plus placebo first, then spironolactone 50 mg QD
Period: Overall Study
Arm/Group | AMB + Spiro First, Then Placebo, Cardiopulmonary Fitness | AMB + Placebo First, Then Spironolactone
Started (First ambrisentan 5 or 10 mg QD + Spiro 50 mg QD (90 d), then washout (21 d), then +placebo (90 d)) | 0 | 2 (Ambrisentan 5 or 10 mg QD + placebo (90 d) first, then washout (21 d), then +Spiro 50 mg QD (90 d).)
Completed | 0 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- AMB + Spiro, Cardiopulmonary Fitness: Ambrisentan 5 or 10 mg every day (QD) Spironolactone 50 mg QD
  Ambrisentan plus Spironolactone: Cardiopulmonary fitness
  Cross over design
Arm/Group | AMB + Spiro, Cardiopulmonary Fitness
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 61 [58 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2
Study-Specific Measure [Count of Participants; unit: Participants] | 2

OUTCOME MEASURES:

1. Primary Outcome: Effect of Combination Ambrisentan + Spironolactone on Peak Volume of Oxygen Consumption (pVO2) and Cardiac Output
Description: Study the effect of combination ambrisentan (5-10 mg/d) + spironolactone (50 mg/d) on pVO2 and cardiac output. The pVO2 refers to a measure of general physical fitness measured during exercise.
Time Frame: Up to average of 20 min
Population: Data were not reported due to patient privacy considerations owing to low enrollment.
Groups:
- AMB + Placebo First: Ambrisentan 5 or 10 mg QD + placebo
Arm/Group | AMB + Spiro, Cardiopulmonary Fitness | AMB + Placebo First
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | AMB + Spiro, Cardiopulmonary Fitness | Placebo Cardiopulmonary Fitness
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

LIMITATIONS AND CAVEATS:
Poor enrollment, study terminated early

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-24): https://cdn.clinicaltrials.gov/large-docs/94/NCT02253394/Prot_SAP_000.pdf